CLINICAL TRIAL: NCT00030368
Title: A Phase I Study of PS-341 in Combination With Paclitaxel in Metastatic Solid Tumors
Brief Title: Bortezomib and Paclitaxel in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01408; 0158; NCI-1857; CDR0000069159; OSU-01H0147; U01CA076576 (NIH)
Record Dates: First submitted 2002-02-14; First posted 2003-04-09 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib; Paclitaxel; Taxes

ARMS (1):
- Treatment (bortezomib, paclitaxel) (Experimental): Patients receive bortezomib IV on days 2 and 9 and paclitaxel IV over 1 hour on days 1 and 8. For the first course only, patients do not receive paclitaxel on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: paclitaxel; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of combining bortezomib with paclitaxel in treating patients who have advanced or metastatic solid tumors. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining bortezomib with paclitaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of bortezomib when given in combination with paclitaxel in patients with locally advanced or metastatic solid tumors.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib.

Patients receive bortezomib IV on days 2 and 9 and paclitaxel IV over 1 hour on days 1 and 8. For the first course only, patients do not receive paclitaxel on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity or greater than 80% 20S proteasome inhibition. Once the MTD is determined, an additional 6-9 patients are accrued and treated at that dose.

Patients are followed at 21 days.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumor for which there is no curative treatment
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)
* Creatinine no greater than ULN
* Left ventricular function at least lower limit of normal if received prior doxorubicin
* No grade II or IV tilt-table test
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No thrombotic event within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction to compounds of similar chemical or biological composition to study drugs
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* Prior paclitaxel allowed
* At least 2 weeks since prior hormonal therapy
* No concurrent steroids or hormonal therapy except steroids to prevent hypersensitivity reactions to paclitaxel or hormonal therapy for non-disease-related conditions (e.g., insulin for diabetes)
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior surgery
* Recovered from prior therapy
* No other concurrent investigational agents
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No concurrent anticoagulation therapy
* Concurrent pamidronate or zoledronate allowed for treatment of hypercalcemia or for palliation of skeletal metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-11; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined as Common Terminology Criteria (CTC) version 2.0 grade 3 or greater non-hematologic toxicity or grade 4 hematologic toxicity with the exception of asymptomatic neutropenia [ANC < 500] | 21 days
Maximum-tolerated dose (MTD) based on the incidence of DLT | 21 days
Dose of PS-341 that results in not more than 70% to 80% 20S proteasome inhibition [20S-PI] in combination with a paclitaxel | At baseline and at 1 hour of weeks 1, 2 and 4

SECONDARY OUTCOMES:
Response according to the Response Evaluation Criteria in Solid Tumors (RECIST) Committee | Up to 21 days
  Reported descriptively using all eligible patients and evaluable patients separately. Response rates will include 95% confidence limits.
Change in the level of p27 and Bax proteins in peripheral blood mononuclear cells | From baseline to 6 hours of day 1 (week 1) and day 2 (week 2)
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.
Change in plasma levels of TNF, IL-1, IL-6, and C-reactive protein | From baseline to 6 hours of day 2 (weeks 1 and 2)
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.
Change in NF-kb biomarkers TRAP I and c-IAP-2 in tumor tissue blocks | From baseline to 6 hours of day 2 (weeks 1 and 2)
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.
Change in phosphorylation of c-Jun and JNK in tumor tissue blocks | From baseline to 6 hours of day 2 (weeks 1 and 2)
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Shapiro, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States